CLINICAL TRIAL: NCT03459599
Title: Antibiotic Prophylaxis in Ragged Placental Membranes: A Prospective, Multicenter, Randomized Trial
Brief Title: Antibiotic Prophylaxis in Ragged Placental Membranes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sarawak General Hospital (Other)
Collaborators: University Malaysia Sarawak (Other)
Responsible Party: Principal Investigator, Voon Hian Yan, Principal Investigator, Sarawak General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16-1016-31034
Record Dates: First submitted 2018-02-23; First posted 2018-03-09 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Endometritis Postpartum; Endometritis; Membranes; Retained
Keywords: Antibiotic; Endometritis; Placental membranes; Prophylaxis; Ragged membranes
MeSH Terms: conditions — Endometritis | interventions — Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylaxis (Active Comparator): Current protocol of administering antibiotics maintained
  Interventions: Drug: Prophylactic antibiotics
- No prophylaxis (Active Comparator): Antibiotics withheld, with appropriate observation and follow up
  Interventions: Other: No prophylaxis (Amox-clav withheld)

INTERVENTIONS:
Drug: Prophylactic antibiotics — Amox-clav given to eligible women as per existing protocol, which is 625mg three times a day, for a week
  Other Names: Amox-clav given as per protocol
  Arms: Prophylaxis
Other: No prophylaxis (Amox-clav withheld) — Withholding Amox-clav, which is the current local practice for women with ragged placental membranes. This was replaced with appropriate counselling on signs and symptoms of endometritis, when and where women should present if the symptoms above occur. A follow up phone call was performed at 2 weeks and 6 weeks postpartum to ascertain well-being of patients
  Other Names: Expectant management
  Arms: No prophylaxis

SUMMARY:
In some centres, women are routinely given a course of antibiotics postnatally if ragged placental membranes were present at delivery. The investigators examined the necessity such an intervention.

DETAILED DESCRIPTION:
Postpartum endometritis resulting in sepsis remain one of the leading cause of maternal mortality in developing countries. Ragged placental membrane is a risk factor for endometritis and is not infrequently encountered. Several hospitals in Malaysia, largely those geographically-removed currently practice administering prophylactic antibiotics for women with ragged placental membranes. The aim is to reduce the risk of postpartum endometritis in a subgroup of women who may present in dire straits. The investigators sought to examine the necessity of such protocols.

ELIGIBILITY:
Inclusion Criteria:

All women who delivered vaginally beyond 24+0 weeks of gestation and were found to have ragged or retained placental membranes immediately after the third stage of labour were invited to participate in the study.

Exclusion Criteria:

1. Fever, within 5 days preceding delivery (Axillary temperature > 37.5oC on 2 or more occasions at least 1 hour apart or temperature > 38oC on one occasion). This also includes intrapartum fever.
2. Required oral or intravenous antibiotics for any other obstetric-related (ex. third or fourth degree tears, preterm prelabour rupture of membranes) or non- obstetric related (ex. pneumonia, acute pyelonephritis) reasons
3. Prolonged rupture of membrane (>18 hours)
4. Retroviral disease, on long term oral or parenteral steroid or receiving other forms of immunosuppressants, including chemotherapy within the last one year.
5. Vaginal delivery for an intrauterine death
6. Penicillin allergy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 716 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Incidence of postpartum endometritis | 6 weeks postpartum
  Postpartum endometritis is defined as follows, when presenting anytime within 6 weeks postpartum
  1. Fever (Axillary temperature > 37.5 degrees Celcius on 2 or more occasions at least 1 hour apart or temperature > 38 degrees Celcius on one occasion), occurring in the absence of apparent source of infection or alternative foci of infection.
  2. Increasing lochia loss or offensive lochia.
  3. Lower abdominal pain or suprapubic tenderness on palpation.
  The diagnosis is further supported by the following:
  1. Elevated total white cell count > 11.0 x 109 cells/L
  2. Positive genital swab culture.
  Incidence is calculated as follows:
  Number of patients diagnosed with endometritis in each arm/total number of patients allocated to each arm

SECONDARY OUTCOMES:
ICU admission rate | 6 weeks postpartum
  ICU admission as a result of endometritis. It is measured as follows:
  a. ICU admission rate in prophylactic antibiotic group= (Number of patients requiring ICU admissions and given antibiotic prophylaxis, regardless of duration/total number of patients given antibiotics prophylaxis )
  a. ICU admission rate in "no prophylaxis" group
  = (Number of patients requiring ICU admissions and NOT given antibiotic prophylaxis, regardless of duration/total number of patients NOT given antibiotics prophylaxis)
Rate of surgical evacuation of retained products of conception | 6 weeks postpartum
  Surgical procedure required as a result of ragged placental membrane or its complications. It is calculated as follows
  1. Surgical evacuation of retained products of conception in prophylaxis group= (Number of patients requiring surgical procedure and given antibiotic prophylaxis, regardless of duration/total number of patients given antibiotics prophylaxis )
  2. Surgical evacuation of retained products of conception in "no prophylaxis" group= (Number of patients requiring surgical procedure and NOT given antibiotic prophylaxis, regardless of duration/total number of patients NOT given antibiotics prophylaxis )
Rate of Blood transfusion | 6 weeks postpartum
  Pack cell transfusion required as secondary to a complication from ragged placental membranes. This can be due to postpartum endometritis or surgical evacuation. It is calculated based on the number of patients requiring transfusion. The number of pack cells required per patient would be also be described.
  1. Blood transfusion in prophylaxis group= (Number of patients requiring pack cell transfusion and given antibiotic prophylaxis, regardless of duration/total number of patients given antibiotics prophylaxis )
  2. Blood transfusion in "no prophylaxis group"= (Number of patients requiring pack cell transfusion and were NOT given antibiotic prophylaxis, regardless of duration/total number of patients NOT given antibiotics prophylaxis )

CONTACTS AND LOCATIONS:
Overall Officials: Hian Yan Voon, MRCOG, Principal Investigator — Sarawak General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meaney-Delman D, Bartlett LA, Gravett MG, Jamieson DJ. Oral and intramuscular treatment options for early postpartum endometritis in low-resource settings: a systematic review. Obstet Gynecol. 2015 Apr;125(4):789-800. doi: 10.1097/AOG.0000000000000732. PMID 25751198
- [Background] Newton ER, Prihoda TJ, Gibbs RS. A clinical and microbiologic analysis of risk factors for puerperal endometritis. Obstet Gynecol. 1990 Mar;75(3 Pt 1):402-6. PMID 2406660
- [Background] van Schalkwyk J, Van Eyk N; INFECTIOUS DISEASES COMMITTEE. Antibiotic prophylaxis in obstetric procedures. J Obstet Gynaecol Can. 2010 Sep;32(9):878-884. doi: 10.1016/S1701-2163(16)34662-X. PMID 21050523
- [Background] Chongsomchai C, Lumbiganon P, Laopaiboon M. Prophylactic antibiotics for manual removal of retained placenta in vaginal birth. Cochrane Database Syst Rev. 2014 Oct 20;2014(10):CD004904. doi: 10.1002/14651858.CD004904.pub3. PMID 25327508
- [Background] Chibueze EC, Parsons AJ, Ota E, Swa T, Oladapo OT, Mori R. Prophylactic antibiotics for manual removal of retained placenta during vaginal birth: a systematic review of observational studies and meta-analysis. BMC Pregnancy Childbirth. 2015 Nov 26;15:313. doi: 10.1186/s12884-015-0752-4. PMID 26610697
- [Background] Fernandez H, Gagnepain A, Bourget P, Peray P, Frydman R, Papiernik E, Daures JP. Antibiotic prophylaxis against postpartum endometritis after vaginal delivery: a prospective randomized comparison between Amox-CA (Augmentin) and abstention. Eur J Obstet Gynecol Reprod Biol. 1993 Aug;50(3):169-75. doi: 10.1016/0028-2243(93)90197-k. PMID 8262292
- [Derived] Voon HY, Pow JY, Tan LN, Suharjono HN, Teo WS. Antibiotic prophylaxis in ragged placental membranes: a prospective, multicentre, randomized trial. BMC Pregnancy Childbirth. 2019 Jul 11;19(1):240. doi: 10.1186/s12884-019-2373-9. PMID 31296180